CLINICAL TRIAL: NCT07128225
Title: Health-related Quality of Life, Electrocardiographic and Holter Findings in Children With Familial Mediterranean Fever
Status: Active, not recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Safaa Kamel Ahmed, Pediatric Specialist, Sohag University
Other Study IDs: Soh-MED-25-6-1MD
Record Dates: First submitted 2025-08-11; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Familial Mediterranean Fever
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Familial Mediterranean fever (FMF) also known as 'periodic peritonitis,' 'familial paroxysmal polyserositis,' 'periodic disease,' 'Siegal-Cattan-Mamou disease,' 'Wolff periodic disease' or 'Reimann syndrome' is an autosomal recessive autoinflammatory disease that causes recurrent fevers and serositis. FMF is caused by a mutation in the Mediterranean fever (MEFV) gene located on the short arm of chromosome 16. This gene produces a protein called pyrin which binds to an apoptosis-associated speck-like protein (ASC) and caspase-1 to inhibit activation of IL-1beta (interleukin) and hence, the inflammatory pathways. Mutation of MEFV genes disrupts pyrin protein and its function, which leads to activation of IL-1beta and then the entire inflammatory pathway.

FMF affects primarily the populations located on the Mediterranean basin mainly Armenians, Turks, Arabs and non-Ashkenazi Jews. However, some new cases have been described in European countries. Turkey is presumed the country with the highest number of FMF patients worldwide, with a prevalence ranging from 1:400 to 1:1000. The exact prevalence of FMF among Arab countries is unknown.

FMF manifests as recurrent attacks of fever and serositis causing severe chest, abdominal, or joint pain. Erysipelas like lesions, scrotal swelling and myalgia can also occur. Patients feel normal between attacks. The severity of the attacks may vary each time, and the time between two attacks could be anywhere from one week to even several years. Some patients reported particular triggers with the appearance of attacks like severe stress, cold exposure, heavy exercise, recent infection, recent surgery, and menstruation. The first attack frequently occurs in childhood, and it usually begins before the age of 20 years. All attacks develop over 2 to 4 hours and last anywhere from 6 hours to 4 days. Colchicine has been the treatment of choice for this disease since 1972.

Amyloidosis is the most common complication of FMF, determining whether the prognosis of the disease is associated with progression to nephrotic syndrome and end-stage renal disease. Colchicine prevents the occurrence of amyloidosis, to stop amyloidosis, and even regress it. The duration of the disease is not the main cause of amyloidosis but specific genetic and environmental conditions is necessary. Early atherosclerosis, ankylosing spondylitis and peritoneal mesothelioma due to chronic inflammation were also reported.

WHO (1997) defined quality of life (QoL) as someone's perception of his position in life depending on the cultural environment, his goals, expectations, principles and values. It is a multidimensional concept, encompasses individuals' physical, emotional health, psychological state, level of independence, social achievements and spiritual state. QoL is dynamic; its perception changes with changing priorities and beliefs of the individual (5). Health related quality of life (HRQoL) is the effect of medical disorder or treatment on individual's physical, emotional, and social well-being. The HRQoL measurement therefore attempts to capture QoL in the context of one's health and illness. In addition, HRQoL also involves an individual's satisfaction about his life, general health and well-being.

WHO declared that the goal of treatment not merely to decrease symptoms and improve signs but also to improve patient's HRQoL. HRQoL has been progressively acknowledged as an essential outcome measure in clinical trials and health service research and evaluation. It is essential to evaluate QoL to clearly understand the effects of diseases on children to help making decisions and adjust plans. Moreover, improving the QoL in children and adolescents with chronic diseases is a very important long-term goal in paediatric rehabilitation.

Thomas and colleagues in their research studied HRQoL of 118 children with FMF and 100 healthy controls in Cairo using PedsQL 4.0 Generic Core Scale and illustrated that HRQoL was significantly lower in FMF compared to healthy controls (mean ± SD of total score was 33.97 ± 12.61 and 85.29 ± 14.03, for diseased and control group respectively, P value: <0.001). Also, HRQoL total score was significantly negatively correlated with frequency of the attacks (r = -.49, P value: <0.001) and with disease severity (r = -0.74, P value: <0.001). (8) Cardiovascular system involvement is among the causes of high morbidity and mortality in FMF. Different cardiovascular complications had been reported in FMF as valvular affection, pericarditis, pericardial effusion, cardiomyopathy and ventricular dysfunction were reported among patients with FMF. FMF causes also variations in the duration of the action potential creating cardiac repolarization abnormalities causing arrhythmias even without the presence of amyloidosis and can occur' not only during periods of attack but also in patients who do not experience attack. (9) Cardiac autonomic nervous system (ANS) plays an integral

DETAILED DESCRIPTION:
Familial Mediterranean fever (FMF) also known as 'periodic peritonitis,' 'familial paroxysmal polyserositis,' 'periodic disease,' 'Siegal-Cattan-Mamou disease,' 'Wolff periodic disease' or 'Reimann syndrome' is an autosomal recessive autoinflammatory disease that causes recurrent fevers and serositis. FMF is caused by a mutation in the Mediterranean fever (MEFV) gene located on the short arm of chromosome 16. This gene produces a protein called pyrin which binds to an apoptosis-associated speck-like protein (ASC) and caspase-1 to inhibit activation of IL-1beta (interleukin) and hence, the inflammatory pathways. Mutation of MEFV genes disrupts pyrin protein and its function, which leads to activation of IL-1beta and then the entire inflammatory pathway. (1) FMF affects primarily the populations located on the Mediterranean basin mainly Armenians, Turks, Arabs and non-Ashkenazi Jews. However, some new cases have been described in European countries. Turkey is presumed the country with the highest number of FMF patients worldwide, with a prevalence ranging from 1:400 to 1:1000. The exact prevalence of FMF among Arab countries is unknown. (2) FMF manifests as recurrent attacks of fever and serositis causing severe chest, abdominal, or joint pain. Erysipelas like lesions, scrotal swelling and myalgia can also occur. Patients feel normal between attacks. The severity of the attacks may vary each time, and the time between two attacks could be anywhere from one week to even several years. Some patients reported particular triggers with the appearance of attacks like severe stress, cold exposure, heavy exercise, recent infection, recent surgery, and menstruation. The first attack frequently occurs in childhood, and it usually begins before the age of 20 years. All attacks develop over 2 to 4 hours and last anywhere from 6 hours to 4 days. Colchicine has been the treatment of choice for this disease since 1972. (3) Amyloidosis is the most common complication of FMF, determining whether the prognosis of the disease is associated with progression to nephrotic syndrome and end-stage renal disease. Colchicine prevents the occurrence of amyloidosis, to stop amyloidosis, and even regress it. The duration of the disease is not the main cause of amyloidosis but specific genetic and environmental conditions is necessary. Early atherosclerosis, ankylosing spondylitis and peritoneal mesothelioma due to chronic inflammation were also reported. (4) WHO (1997) defined quality of life (QoL) as someone's perception of his position in life depending on the cultural environment, his goals, expectations, principles and values. It is a multidimensional concept, encompasses individuals' physical, emotional health, psychological state, level of independence, social achievements and spiritual state. QoL is dynamic; its perception changes with changing priorities and beliefs of the individual (5). Health related quality of life (HRQoL) is the effect of medical disorder or treatment on individual's physical, emotional, and social well-being. The HRQoL measurement therefore attempts to capture QoL in the context of one's health and illness. In addition, HRQoL also involves an individual's satisfaction about his life, general health and well-being. (6) WHO declared that the goal of treatment not merely to decrease symptoms and improve signs but also to improve patient's HRQoL. HRQoL has been progressively acknowledged as an essential outcome measure in clinical trials and health service research and evaluation. It is essential to evaluate QoL to clearly understand the effects of diseases on children to help making decisions and adjust plans. Moreover, improving the QoL in children and adolescents with chronic diseases is a very important long-term goal in paediatric rehabilitation. (7) Thomas and colleagues in their research studied HRQoL of 118 children with FMF and 100 healthy controls in Cairo using PedsQL 4.0 Generic Core Scale and illustrated that HRQoL was significantly lower in FMF compared to healthy controls (mean ± SD of total score was 33.97 ± 12.61 and 85.29 ± 14.03, for diseased and control group respectively, P value: <0.001). Also, HRQoL total score was significantly negatively correlated with frequency of the attacks (r = -.49, P value: <0.001) and with disease severity (r = -0.74, P value: <0.001). (8) Cardiovascular system involvement is among the causes of high morbidity and mortality in FMF. Different cardiovascular complications had been reported in FMF as valvular affection, pericarditis, pericardial effusion, cardiomyopathy and ventricular dysfunction were reported among patients with FMF. FMF causes also variations in the duration of the action potential creating cardiac repolarization abnormalities causing arrhythmias even without the presence of amyloidosis and can occur' not only during periods of attack but also in patients who do not experience attack. (9) Cardiac autonomic nervous system (ANS) plays an integral role in the modulation of normal cardiac electrophysiology and regulating cardiac activity. Abnormalities in the autonomic tone are potentially associated with worse prognosis including life threatening ventricular arrhythmias and sudden cardiac death (SCD). Several studies reported the potential role of ANS in autoimmune rheumatic disorders such as lupus, rheumatoid arthritis and systemic sclerosis. It is suggested that the abnormal autonomic activity in FMF is similar to dysautonomia described in a variety of rheumatic disorders. The status of cardiac ANS can be assessed by various non-invasive methods as heart rate variability (HRV). Canpolat et al reported that patients with FMF showed delayed recovery of heart rate and abnormal HRV and with respect to normal subjects. Cardiac autonomic dysfunctions might be involved in FMF patients even in patients without cardiac symptoms. (10) The risk of cardiac arrhythmias can be predicted from the electrocardiogram (ECG) by measuring several repolarization markers. Some of the most used predictors in clinical practice are: the T wave, QT interval and its correction by heart rate (QTc), QT interval dispersion (QTd), Q wave dispersion and P wave dispersion. (11) Aim of the work

1. To assess HRQoL of FMF children in comparison to healthy controls.
2. To detect ECG, Holter findings and HRV among FMF children in comparison to healthy controls to assess their susceptibility to cardiac repolarization abnormalities and therefore arrhythmia and to detect association between the findings and genetic mutations and treatment of FMF.

Patients and methods Study design Case control study Study setting and duration the study sample will compose of children with FMF and healthy controls admitted at Paediatric Department or attending outpatient Paediatric clinic at Sohag University Hospitals, from protocol acceptance till end of the study.

Study population

* Children with FMF Inclusion criteria

  1. Children diagnosed with FMF and their disease severity was assessed using Tel-Hashomer criteria and the international severity score for FMF (ISSF) (12, 13)
  2. Children below 18 years old
  3. During the attack and in attack-free period for at least 2 weeks
  4. Parents' acceptance for participations
  5. Patients and their parents accepted to answer all the questions of the questionnaire Exclusion criteria

  <!-- -->

  1. Other autoimmune, autoinflammatory, congenital or acquired cardiac diseases, acute or chronic infection.
  2. Parents' refusal for participations
  3. Those who didn't fulfil the inclusion criteria
* Control group The control group will consist of children matching cases in age and gender, with no acute or chronic illnesses, attending Paediatric Outpatient clinic for routine follow up after their parents' consent to participate and the children and their parents accepted to answer all questions of the questionnaire.

Study Tools In order to collect the necessary information for the study, the following data and investigations will be conducted I. History Age Gender Residence School age Mother age Father age Mother education Father education Mother work Father work Age at diagnosis Disease duration Number of attacks per month and per year Hospital admission times Treatment Dose Duration of treatment II. Examination Blood pressure Body surface area Disease severity using ISSF III. Electrocardiogram (ECG): ECG will be carried out for all patients and controls. The following parameters will be measured

1. Axis
2. R-R distance
3. Rhythm
4. QRS voltage
5. T wave measurement
6. PR interval
7. QRS interval
8. QT interval: was measured manually from the point where the Q wave started and the T wave returned to the isoelectric line.
9. QT dispersion: were defined as the difference between the longest and shortest QT.
10. Corrected QT (QTc): were performed with the Bazett's formula QTc = QT / √RR Where QTc is the corrected QT interval, QT interval is the distance from Q wave to end of T wave and RR is the time from two consecutive R waves.

IV. Holter ambulatory Electrocardiogram monitoring

* Duration: 24 hours.
* Type of machine: Mortara 2016 american made H3+.
* Software: Mortara Company American made.
* Holter monitoring will be applied to all children, minimum, mean, maximum heart rate, rhythms, corrected QT by Bazett's formula and heart rate variability will be evaluated.

V. PedsQL4.0 Generic Core Scales The PedsQL4.0 scale is a validated questionnaire developed by Varni et, al to assess the HRQOL in children (cases and control), includes 21 items for 2-4 years and 23 items for all other age groups. It comprises child report (5-18 years of age) and parent report (2-18 years of age) of the child's HRQOL. The PedsQL assesses physical (8items), emotional (5items), social (5items) and school/nursery school (5/3 items) functioning in adolescents and children. For children 8-18 years of age and parent/proxy report formats. The pediatric forms (including ages 5-7 years, 8-12 years, and 13-18 year), filled in by children, and parental forms (including ages 2-4, 5-7, 8-12, 13-18 years), filled in by their parents. Items are rated on a 5-point ordinal scale to indicate the problems children encounter in various areas of functioning, ranging from 0 (never) to 4 (almost always). For younger children, the ordinal scale is reworded and simplified to a 3-point scale: 0 (not at all a problem), 2 (sometimes a problem) and 4 (a lot of problem). From the sum of the raw scores from the 23 (or 21) items, a summary score ranging from 0 to 100 can be calculated, with higher scores indicating higher. (14) Confidentiality and ethical consideration

1. Approval of the concerned administrative authority (Medical Research Ethics Committee of Sohag University) will be obtained
2. Written informed consent after explaining the aim of the study will be obtained from parents of children of both groups who will participate in the study.
3. The questionnaire used in data collection will be anonymous and confidentiality of responses will be assured.

ELIGIBILITY:
Inclusion Criteria:

* 1. Children diagnosed with FMF and their disease severity was assessed using Tel-Hashomer criteria and the international severity score for FMF (ISSF) (12, 13) 2. Children below 18 years old 3. During the attack and in attack-free period for at least 2 weeks 4. Parents' acceptance for participations 5. Patients and their parents accepted to answer all the questions of the questionnaire

Exclusion Criteria:

Exclusion criteria

1. Other autoimmune, autoinflammatory, congenital or acquired cardiac diseases, acute or chronic infection.
2. Parents' refusal for participations
3. Those who didn't fulfil the inclusion criteria -

Ages: 5 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: the study sample will compose of children with FMF and healthy controls admitted at Paediatric Department or attending outpatient Paediatric clinic at Sohag University Hospitals, from protocol acceptance till end of the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
QT interval | one year
  QT interval represents the total time it takes for the ventricles to depolarize and then repolarize

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospitals, Sohag, Egypt

REFERENCES:
- [Background] Bhatt H, Cascella M. Familial Mediterranean Fever. 2023 Jul 31. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK560754/ PMID 32809589
- [Background] Bodur H, Gul Yurdakul F, Duruoz MT, Cay HF, Ucar U, Keskin Y, Sargin B, Gurer G, Yurdakul OV, Calis M, Deveci H, Aydin Y, Hizmetli S, Cevik R, Karahan AY, Ataman S, Ecesoy H, Gunendi Z, Toprak M, Sen N, Altintas D, Cengiz AK, Caglayan G, Demir AN, Kaplan H, Ketenci S, Melikoglu MA, Nayimoglu M, Nas K, Sarifakioglu B, Sezer I. Familial Mediterranean fever: Health-related quality of life and associated variables in a national cohort. Arch Rheumatol. 2020 Dec 10;36(2):159-166. doi: 10.46497/ArchRheumatol.2021.8215. eCollection 2021 Jun. PMID 34527919
- [Background] Martin MP, McEntee ML, Suri Y. Caregiver Quality of Life: How to Measure It and Why. Am J Health Promot. 2021 Sep;35(7):1042-1045. doi: 10.1177/08901171211030142f. No abstract available. PMID 34351244
- [Background] Assouad E, El Hage S, Safi S, El Kareh A, Mokled E, Salameh P. Familial Mediterranean fever research activity in the Arab world: the need for regional and international collaborations. East Mediterr Health J. 2021 Oct 27;27(10):984-992. doi: 10.26719/emhj.21.036. PMID 34766324